CLINICAL TRIAL: NCT05913089
Title: A Phase II/III Clinical Study on the Efficacy and Safety of TQB2450 Injection Combined With Chemotherapy or Anlotinib Hydrochloride Capsule in the Perioperative Treatment of Resectable Stage II/III Non Small Cell Lung Cancer.
Brief Title: A Clinical Study of TQB2450 Injection Combined With Chemotherapy or Anlotinib Hydrochloride Capsule in the Treatment of Non Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-II/III-01
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2022-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2450 injection + Chemotherapy (Experimental): TQB2450 injection combined with chemotherapy, 21 days as a treatment cycle.
  Interventions: Drug: TQB2450 injection + Chemotherapy
- TQB2450 injection + Anlotinib Hydrochloride Capsule (Experimental): TQB2450 injection combined with anlotinib hydrochloride capsule, 21 days as a treatment cycle.
  Interventions: Drug: TQB2450 injection + Anlotinib Hydrochloride Capsule

INTERVENTIONS:
Drug: TQB2450 injection + Chemotherapy — TQB2450 injection is a humanized monoclonal antibody targeting programmed death ligand -1 (PD-L1).
  Chemotherapy is a systematic treatment that kill fast growing cells.
  Arms: TQB2450 injection + Chemotherapy
Drug: TQB2450 injection + Anlotinib Hydrochloride Capsule — TQB2450 injection is a humanized monoclonal antibody targeting programmed death ligand -1 (PD-L1).
  Anlotinib hydrochloride is a muti-target tyrosine kinase inhibitor.
  Arms: TQB2450 injection + Anlotinib Hydrochloride Capsule

SUMMARY:
This is a clinical study on the efficacy and safety of TQB2450 injection combined with chemotherapy or anlotinib hydrochloride capsule in the perioperative treatment of resectable non-small cell lung cancer. The part I study was planned to enroll 58 subjects, 1:1 randomized into two cohorts. The treatment regimen was as follows: Cohort 1: 3-4 cycles of TQB2450 combined with chemotherapy, surgery should be performed 4-6 weeks after the last administration, and TQB2450 therapy should be continued for 1 year after surgery. Cohort 2: 4 cycles of TQB2450 combined with 3 cycles of anlotinib hydrochloride capsule. Surgery was performed 4-6 weeks after the last dose and continued for 1 year starting 4 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients with stage II-IIIB (T3N2M0 only) Non-Small Cell Lung Carcinoma (NSCLC) and determined to be eligible for curable R0 excision, after pathologic diagnosis of puncture specimens;
* ≥18 years old (calculated on the date of signing the informed consent); Both men and women; Eastern Cooperative Oncology Group (ECOG) score 0~1; Predicted survival ≥3 months;
* Have at least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 criteria within 28 days prior to initiation of treatment;
* Has not received systemic antitumor therapy, including radiotherapy, chemotherapy and immunotherapy;
* Agree to provide fresh or 6 month tumor tissue for programmed death ligand -1 (PD-L1) testing.
* Major organs are functioning well.
* Women of reproductive age should agree that they must use effective birth control during the study period and for 6 months after the study, and that a negative serum or urine pregnancy test occurred within 7 days prior to study enrollment; Men should agree that effective contraception must be used during the study period and for 6 months after the study period ends.
* The subjects voluntarily joined the study and signed the informed consent with good compliance.

Exclusion Criteria:

* Present or complication with other malignancies within 5 years.
* Subjects are known to have genetic abnormalities with approved targeted drug therapy.
* Cirrhosis, active hepatitis;
* Cardio-cerebrovascular abnormalities;
* Subjects with severe active infection within 4 weeks prior to initiation of study treatment; Or unexplained fever >38.0 ℃ occurred during screening and before first administration;
* Patients with active tuberculosis within 1 year prior to enrollment;
* Immunodeficiency disease;
* History of active autoimmune disease or autoimmune disease;
* Preparing for or having previously received an organ transplant, or having received a hematopoietic stem cell transplant within 60 days prior to initial medication, or having a significant host transplant response;
* Patients who required immunosuppressive, systemic, or absorbable topical hormone therapy for immunosuppressive purposes and continued use within two weeks prior to randomization
* Severe infection of grade 4 or higher occurred within 1 year prior to initiation of study therapy;
* Severe lung disease;
* History of pituitary or adrenal dysfunction;
* History of severe mental disorder;
* History of drug abuse, alcoholism or drug use;
* Participated in clinical trials of other drugs within 30 days;
* History of live attenuated vaccine vaccination within 28 days prior to randomization or planned live attenuated vaccine vaccination during the study period;
* Received Chinese patent drugs with anti-tumor indications specified in the National Medical Product Administration approved drug package inserts within 2 weeks prior to initiation of administration
* Had major surgery within 4 weeks prior to initiation of medication;
* Other severe, acute, or chronic medical conditions or laboratory abnormalities that, in the investigator's opinion, may increase the risks associated with study participation or may interfere with the interpretation of the study results, or are otherwise unsuitable for participation in the clinical study;
* The compliance of patients to participate in this clinical study is estimated to be insufficient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) | Baseline up to 60 months.
  MPR defined as the percentage of subjects with a residual surviving tumor less than or equal to 10% after surgery.

SECONDARY OUTCOMES:
Overall survival (OS) | Baseline up to 60 months.
  From randomization to the time of death from any cause.
2/3 year OS rate | Baseline up to 36 months.
  The ratio of two-year survival to three-year survival.
Event free survival (EFS) assessed by the investigator. | Baseline up to 60 months.
  From the time of randomization to the occurrence of a predetermined event, including death, disease progression, change to chemotherapy, change to chemotherapy, addition of other treatments, occurrence of fatal or intolerable side effects, etc.
Disease free survival (DFS) assessed by Blinded Independent Central Review (BICR) | Baseline up to 60 months.
  The time from randomization to the onset of tumor recurrence or death from any cause.
Pathological complete response (pCR) | Baseline up to 4 months.
  Ratio of patients with no residual cancer cells found in the pathological examination after treatment.
R0 resection rate | Baseline up to 4 months.
  The proportion of subjects who could undergo R0 resection, which is one of the surgery-related end points.
Surgical delay rate | Baseline up to 4 months.
  The proportion of subjects who could not undergo surgery in time after neoadjuvant therapy.
Pathological downgrading rate | Baseline up to 4 months.
  The proportion of patients with reduced lung cancer stage determined by pathological results after surgery.

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Cancer Hospital of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Weifang People's Hospital, Weifang, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality